CLINICAL TRIAL: NCT04214990
Title: Effect of Low-dose Aspirin for Stomach Cancer Prevention After Endoscopic Resection of Gastric Neoplasm (EASTERN): a Randomized Controlled Trial
Brief Title: Aspirin Use for Gastric Cancer Prevention in the Early Gastric Cancer Patients
Acronym: EASTERN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Incheon St.Mary's Hospital/The Catholic University (Unknown); Kosin University Gospel Hospital (Other); Pusan National University Hospital (Other); SMG-SNU Boramae Medical Center (Other); Chonnam National University Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Chilgok Kyungpook National University (Unknown); Hallym University Medical Center (Other); Asan Medical Center (Other); Seoul National University Bundang Hospital (Other); Severance Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Il Ju Choi, Gastroenterologist, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCC2019-0184
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Aspirin; Gastric Cancer
Keywords: Aspirin; Gastric cancer prevention; Endoscopic submucosal dissection
MeSH Terms: conditions — Stomach Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Active Comparator): Enteric coated aspirin
  Interventions: Drug: Aspirin 100mg
- Placebo (Placebo Comparator): Enteric coated aspirin placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Aspirin 100mg — Daily aspirin 100 mg for 5 years
  Arms: Aspirin
Drug: Placebo oral tablet — Daily placebo for 5 years
  Arms: Placebo

SUMMARY:
This study aimed to investigate the effect of low-dose (100 mg) asprin on the prevention of gastric cancer in the early gastric cancer patients with negative H. pylori status who underwent endoscopic submucosal dissection.

DETAILED DESCRIPTION:
Aspirin has been widely used as an anti-platelet drug for the primary or secondary prevention of cardiovascular events, including ischemic heart disease and stroke. In 2016, the U.S. Preventive Services Task Force recommended initiating low-dose aspirin use for the primary prevention of cardiovascular diseases and colorectal cancer in adult aged 50 to 59 years who have a 10% or greater 10-year cardiovascular disease risk, are not at increased risk of bleeding, have a life expectancy of at least 10 years, and are willing to take low-dose aspirin daily for at least 10 years. In addition, a meta-analysis reported that long-term aspirin use was associated with reduced the risk of gastrointestinal cancers including colorectal cancer, esophageal cancer, and gastric cancer. However, most studies that reported the cancer prevention effect of long-term aspirin use were conducted as a secondary analysis or subgroup analysis of primary studies investigating the aspirin use for cardiovascular disease prevention. Thus, there is a limitation that appropriate sample sizes and follow-up periods for the cancer prevention effect of aspirin were not considered.

In 2018, we reported that H. pylori treatment reduced the development of metachronous gastric cancer after endoscopic resection in early gastric cancer patients. However, metachronous gastric cancer could develop after successful H. pylori eradication with an annual incidence of 1%-3%. Therefore, we designed a multi-center, double-blind, randomized, placebo-controlled trial to evaluate whether long-term low-dose (100 mg) aspirin uses prevents gastric cancer in early gastric cancer or high-grade dysplasia patients who underwent endoscopic resection.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 19-70 years who underwent endoscopic resection for high-grade adenoma or early gastric cancer (category 4 [non-invasive high grade neoplasm] or category 5 [invasive neoplasia] according to the Vienna classification of gastrointestinal epithelial neoplasia [Schlemper RJ, et al. Gut 2000;47:251-255.])
* Final pathological results after endoscopic resection met the absolute or expanded criteria according to the Japanese Gastric Cancer Treatment guideline 2014 (version 4)
* Patients who had negative H. pylori status or those who eradicated H. pylori status
* Willingness to sign an informed consent form

Exclusion Criteria:

* Patients who received aspirin for the secondary prevention of cardiovascular diseases or cerebrovascular diseases
* Regular aspirin uses (more than 3 times a week) with 2 months before screening visit
* Patients who used anticoagulants or antiplatelet drugs for therapeutic purpose
* Previous gastrectomy history
* Current treatment for serious medical condition which could hinder participation (such as severe heart dysfunction, liver cirrhosis, renal failure, COPD or bronchial asthma, or uncontrolled infection)
* High risk patients for bleeding complications (cerebral aneurysm, vascular malformation, esophageal or gastric varices, or hemophilia, etc)
* Active peptic ulcer disease (patients who treated peptic ulcer completely could be enrolled)
* Diagnosis and active treatment for other organ cancer (except carcinoma in situ, and non-melanoma skin cancer) within 5 years
* Non-curative resection of early gastric cancer after endoscopic resection
* Aspirin allergy or contraindication of aspirin use
* Pregnant or lactating women
* Alcoholism, drug abuse
* Inadequate patients for study enrollment according to the evaluation of the study physician
* Inability to provide an informed consent
* Patients who took a 28-day run-in-period medication less than 80%

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of gastric cancer between the intervention and placebo groups | Until last enrolled patients take 5-year trial medication
  Histologically confirmed gastric cancer detected at follow-up endoscopy or registered at the Korean Cancer Registry

SECONDARY OUTCOMES:
All-cause mortality | Until last enrolled patients take 5-year trial medication
  Mortality from any causes
The incidence of cardiovascular disease and cerebrovascular disease between the intervention and placebo groups | Until last enrolled patients take 5-year trial medication
  Cardiovascular diseases (stable and unstable angina, myocardial infarction); Cerebrovascular diseases (transient ischemic attack, cerebral infarction, other small vascular infarction, etc)
The incidence of other organ cancers between the intervention and placebo groups | Until last enrolled patients take 5-year trial medication
  Cancers detected at follow-up visits or registered at the Korean Cancer Registry
The incidence of gastric dysplasia (adenoma) between the intervention and placebo groups | Until last enrolled patients take 5-year trial medication
  Histologically confirmed gastric dysplasia (adenoma) detected at follow-up endoscopy
Complication related to the aspirin use | Until last enrolled patients take 5-year trial medication
  Gastrointestinal bleeding, intracranial hemorrhage, subarachnoid hemorrhage, and other bleeding complications
Improvement of atrophy and intestinal metaplasia | At the time of 5-year trial medication
  Change in histologic atrophy and intestinal metaplasia grades from enrollment to subsequent endoscopic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Il Ju Choi, M.D., Ph.D., Study Director — National Cancer Center, Korea
Locations (10):
- South Korea (10):
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang
  - Chonnam National University Hospital, Gwangju
  - Incheon St.Mary's Hospital/The Catholic University, Incheon
  - Chung-Ang University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No